CLINICAL TRIAL: NCT04719377
Title: A Prospective, Multi-center, Open-label, Randomized, Controlled Non-inferiority Clinical Trial Evaluating the Effectiveness and Safety of the PowerMe Midline Catheter Versus Traditional PIV in the Chinese Population
Brief Title: A Clinical Trial Evaluating the Effectiveness and Safety of the PowerMe Midline Catheter in the Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-19POWME01
Record Dates: First submitted 2020-12-28; First posted 2021-01-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Catheterization
Keywords: midline; overall performance; indwelling time

STUDY DESIGN:
Intervention Model Description: PowerMe Midline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powerme midline catheter (Experimental): Powerme midline catheter
  Interventions: Device: catheter placement
- peripheral intravenous catheter (Sham Comparator): BD Pegusas peripheral intravenous catheter
  Interventions: Device: catheter placement

INTERVENTIONS:
Device: catheter placement — catheter placement

SUMMARY:
This study is designed to evaluate the effectiveness and the safety of the PowerMeTM Midline Catheter in the Chinese population.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, randomized, controlled, non-inferiority clinical trial designed to evaluate the effectiveness and the safety of the PowerMeTM Midline Catheter compared to PIVC in the Chinese population in order to support the product's registration in China.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. Inpatient with a need for intravenous infusion for an expected period of more than 4 days but no more than 28 days;
3. The veins in the upper limbs is suitable for puncture and catheterization of both the investigational device and the control device;
4. Willing to provide written Informed Consent and complete the study per the protocol.

Exclusion Criteria:

1. Coagulation disorder or active bleeding;
2. Skin injury, infection, or dermatosis at the site to be punctured;
3. History of radiotherapy, thrombosis, or vascular surgery; arteriovenous fistula or phlebitis history at the area and/or vein to be catheterized;
4. History of mental illness;
5. End stage renal disease requires vein protection;
6. Conditions with decreased venous flow in the extremity, such as lymphedema of the arm, etc.;
7. Infusions of vesicant or irritant drugs, hyperosmotic infusate (the osmotic pressure >900mOsm/L in this study), parenteral nutrition, etc., which are not suitable for peripheral intravenous infusion (If other appropriate venous access is established for the aforementioned infusates, the patient may be enrolled).
8. The evaluation of the upper limb veins is Grade II, the evaluation grade is as following:

   * 0 Veins are obviously bulged on the skin surface. The veins are touchable, thick, straight, soft, elastic and fixed.
   * I Veins are relatively full and faintly touchable. The veins are less elastic or slide easily.
   * II Veins are not full or collapsed and untouchable. The veins are hard or sliding. Phlebitis.
9. Self-reported being pregnant or lactating;
10. Other conditions that the investigator considers improper for the study;
11. Participating in another study or already enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Acceptance of the overall performance of the IV catheter system | up to 28 days
  After the placement of the IV catheter system, the study nurse shall answer "yes/no" to the following questions:
  1. Can the IV catheter system vent the air properly;
  2. Can the IV catheter system be inserted and be placed in the blood vessel;
  3. Can the needle tube be withdrawn from the septum;
     After the removal of the IV catheter system, the study nurse shall answer "yes/no" to the following questions:
  4. Can the IV catheter system be removed properly;
  5. There is no leakage during the application of the IV catheter system (including the processes of venting, infusion, flushing and sealing, and indwelling).

SECONDARY OUTCOMES:
Success rate of the first insertion of the catheter | First day, during catheter insertion
  Successful first insertion means the IV catheter system can be successfully inserted into the blood vessel on the first insertion.
Indwelling time | up to 28 days
  The retention time of the IV catheter system of each subject after successful insertion.
Rate of good performance of the pinch clamp | up to 28 days
  If the pinch clamp can close and open the tubing properly, performance of the pinch clamp can be evaluated as "good".
Incidence of catheter blockage | up to 28 days
  The catheter system is blocked, causing the system to fail to infuse the fluid after it is connected to the infusion set/syringe.
Incidence of accidental dislodgement | up to 28 days
  Unintentional premature removal of the catheter from the vessel.
Incidence of phlebitis | up to 28 days
  Incidence of phlebitis
Incidence of adverse events | up to 28 days
  Incidence of adverse events
Incidence of serious adverse events | up to 28 days
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xuying Li, RN, Principal Investigator — Hunan Cancer Hospital, China
Locations (4):
- China (4):
  - Hunan Cancer Hospital, Changsha
  - Shanghai First General Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No